CLINICAL TRIAL: NCT05718856
Title: A Multicenter, Randomized, Open-label StudyTo Compare The Efficacy And Safety Of TPO-RAs Combining Anti-CD 20 Monoclonal Antibody Versus TPO-RAs in Persistent or Chronic Pediatric ITP Patients Who Failed or Relapse After Glucocorticoid Therapy
Brief Title: TPO-RAs Combining Anti-CD 20 Monoclonal Antibody Versus TPO-RAs in the Management of Pediatric Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Beijing Children's Hospital (Other); Tianjin People's Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Henan Cancer Hospital (Other Government); Tianjin Medical University Second Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022047
Record Dates: First submitted 2022-11-13; First posted 2023-02-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-02

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: immune thrombocytopenia; autoantibody; eltrombopag; rituximab
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- efficacy of TPO-RAs (Active Comparator): After enrollment, all subjects receive TPO-RAs treatment. The initial dose of eltrombopag administration was an oral 37.5 mg (6-11 years old) or 50 mg (12-17 years old) once daily. The initial dose of hetrombopag administration was an oral 3.75 mg (6-11 years old) or 5mg (12-17 years old) once daily in all participants. The initial dose of avatrombopag administration was an oral 10 mg (<30kg) or 20mg (≥30kg) once daily in all participants. Complete blood count including platelet count was done once a week. The dose of TPO-RAs was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count >250×10^9/L, the TPO-RAs will stop until the platelet count <100×10^9/L.
  Efficacy and safety will be evaluated at Week 4, Week 8, Week 12 and Week 24.
  Interventions: Drug: TPO-RAs
- efficacy of TPO-RAs combining anti-CD 20 monoclonal antibody (Experimental): After enrollment, all subjects receive TPO-RAs treatment. The initial dose of eltrombopag, hetrombopag and avatrombopag administration were the same as patients in TPO-RAs monotherapy group. The dose of TPO-RAs was adjusted according to the subject platelet count. Two kinds of anti-CD 20 monoclonal antibody could be used in this study. All subjects receive single dose infusion of rituximab 375 mg/m(2) within 14 days after enrollment. Subjects weighing less than 30kg will be given rituximab 100 mg once a week for four times. Ortuzumab at 1000mg/ dose is also recommended for subjects weighing 45kg or greater. Ps. Participants in the eltrombopag monotherapy group who have platelet count < 20×10^9/L or significant skin and mucosal bleeding at the end of 12 weeks of treatment will be given a single dose of rituximab 375mg/m2. Ortuzumab at 1000mg/ dose is also recommended for subjects weighing 45kg or greater. Efficacy and safety will be evaluated at Week 4, Week 8, Week 12 and Week 24.
  Interventions: Drug: TPO-RAs combining anti-CD 20 monoclonal antibody

INTERVENTIONS:
Drug: TPO-RAs — After enrollment, all subjects receive TPO-RAs treatment. The initial dose of eltrombopag, hetrombopag and avatrombopag administration were the same as described in arm description. Complete blood count including platelet count was done once a week. The dose of TPO-RAs was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count >250×10^9/L, the TPO-RAs will stop until the platelet count <100×10^9/L.
  Other Names: TPO-R agonists
  Arms: efficacy of TPO-RAs
Drug: TPO-RAs combining anti-CD 20 monoclonal antibody — After enrollment, all subjects receive TPO-RAs treatment. The initial dose of eltrombopag, hetrombopag and avatrombopag administration were the same as described in arm description.The dose of TPO-RAs was adjusted according to the subject platelet count during the period from week 1 to week 24.
  Subjects in TPO-RAs combining anti-CD 20 monoclonal antibody treatment group received single dose infusion of Rituximab 375 mg/m2 within 14 days after enrollment. Subjects weighing less than 30kg will be given Rituximab 100 mg once a week for four times. Ortuzumab at 1000mg/ dose is also recommended for subjects weighing 45kg or greater.
  Ps.Participants in the TPO-RAs monotherapy group who have platelet count < 20×10^9/L or significant skin and mucosal bleeding at the end of 12 weeks of treatment will be given a single dose of Rituximab 375mg/m2 or Ortuzumab at 1000mg/ dose if weighing 45kg or greater.
  Other Names: TPO-R agonist & anti-CD 20 monoclonal antibody
  Arms: efficacy of TPO-RAs combining anti-CD 20 monoclonal antibody

SUMMARY:
This multicenter randomized, open-label study aim to compare the efficacy and safety of TPO-RAs combining anti-CD 20 monoclonal antibody with TPO-RAs in China pediatric ITP patients .This study will be conducted in persistent or chronic pediatric ITP patients who had not responded to or had relapsed after previous glucocorticoid treatment.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the efficacy and safety of TPO-RAs combining anti-CD 20 monoclonal antibody treating previously treated pediatric ITP patients compared to TPO-RAs. The secondary objective was to evaluate the efficacy of TPO-RAs combining anti-CD 20 monoclonal antibody in pediatric ITP patients with positive autoantibody compared to TPO-RAs.In addition, health-related quality of life (HRQoL) measure was assessed in all participants.

166 eligible subjects were randomized to either TPO-RAs combining anti-CD 20 monoclonal antibody or TPO-RAs treatment in 1:1 ratio. 83 enrolled patients are randomly picked up to take TPO-RAs combining with anti-CD 20 monoclonal antibody at the indicated dose. 83 enrolled patients are randomly picked up to take TPO-RAs at the indicated dose.

Three TPO-RAs could be used in this study, including eltrombopag, hetrombopag and avatrombopag. The initial dose of eltrombopag administration was an oral 37.5 mg (6-11 years old) or 50 mg (12-17 years old) once daily in all participants.

The initial dose of hetrombopag administration was an oral 3.75 mg (6-11 years old) or 5mg (12-17 years old) once daily in all participants. The initial dose of avatrombopag administration was an oral 10 mg (<30kg) or 20mg (≥30kg) once daily in all participants.The dose of TPO-RAs was adjusted according to the subject platelet count during the period from week 1 to week 24.

Two kinds of anti-CD 20 monoclonal antibody could be used in this study, including Rituximab and Ortuzumab.Subjects in TPO-RAs combining anti-CD 20 monoclonal antibody treatment group received single dose infusion of Rituximab 375 mg/m2 within 14 days after enrollment. Subjects weighing less than 30kg will be given Rituximab 100 mg once a week for four times. Ortuzumab at 1000mg/ dose is also recommended for subjects weighing 45kg or greater.

Ps.Participants in the TPO-RAs monotherapy group who have platelet count < 20×10^9/L or significant skin and mucosal bleeding at the end of 12 weeks of treatment will be given a single dose of Rituximab 375mg/m2.Ortuzumab at 1000mg/ dose is also recommended for subjects weighing 45kg or greater.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-17 years old (including both ends), male and female;
2. Patients aged 6-11 years (including values at both ends) were diagnosed with chronic ITP, and patients aged 12-17 years (including values at both ends) were diagnosed with persistent or chronic ITP, with platelet counts less than 20×109/L;
3. Patients did not respond to glucocorticoid therapy or relapsed. Previous ITP treatment may include, but is not limited to, glucocorticoids, immunomodulators (IVIG), azathioprine, danazole, cyclophosphamide and immunomodulators.
4. Treatment for ITP (including but not limited to glucocorticoids, recombinant human thrombopoietin, TPO agonist (TPO-RA), azathioprine, danazole, cyclosporin A, mycophenate) must be completed or dose stabilized before enrollment, and therapeutic dose should not be increased after enrollment (e.g. The glucocorticoid dose should be stable for ≥14 days and the immunosuppressant dose should be stable for > 3 months before the first administration of the study drug. TPO drugs should be stopped > 1 month, TPO-RA drugs should be stopped > 1 month).
5. No infectious fever (including but not limited to lung infection) in the past 1 month.
6. Laboratory examination of coagulation function should show that the prothrombin time (PT) and activated partial thrombin time (aPTT) values did not exceed 20% of the normal laboratory value range; No history of abnormal coagulation except for ITP.
7. WBC count, neutrophil absolute value and hemoglobin should be within the normal range of laboratory values. No other abnormality except for ITP. Other exceptions except the following:

   * If the anemia is clearly caused by excessive blood loss associated with ITP.
   * If the increase in WBC count/neutrophil absolute value was clearly due to steroid therapy.
8. Understand the study procedure and voluntarily sign the informed consent.

   * For subjects aged 6-7 (including both ends), parents/guardians understand the study procedure and voluntarily sign the informed consent in person, and subjects are encouraged to participate in the informed process and voluntarily sign the informed consent in person;
   * For subjects aged 8-16 (including both ends), parents/guardians and subjects themselves should understand the study procedure and voluntarily sign the informed consent in person;
   * For the minor subjects > 16 years old, if the subjects rely on their own income as the main source of living, they are regarded as persons with full capacity for civil conduct and can independently carry out legal acts. The subjects can sign informed consent on the premise that they understand the research procedures and are willing to do so;
   * For minor subjects > 16 years old, if the subjects do not rely on their own income as the main source of living, they cannot be regarded as persons with full capacity for civil conduct and cannot independently carry out legal acts. Parents/guardians and subjects should understand the study procedures and voluntarily sign the informed consent in person.

Exclusion Criteria:

1. Subjects who has any history of arterial/venous thrombosis and the following risk factors including clotting factor V Leiden disease, ATIII deficiency, antiphospholipid syndrome, etc..
2. Subjects known to have failed all standard TPO-RAs treatments.
3. Subjects known to have taken anti-CD20 antibodytreatment within 3 months prior to initial use of the study drug.
4. Within 2 weeks prior to the initial use of the study drug, subjects were treated with medications (including but not limited to aspirin, aspirin containing compounds, clopidogrel, salicylate, and/or NSAIDs) or anticoagulants that had an impact on platelet function for > 3 consecutive days.
5. Subjects known to have participated in other investigational clinical trials within 3 months prior to first use of investigational drug.
6. Suffering from severe, progressive, uncontrolled kidney, liver, gastrointestinal, endocrine, lung, heart, nervous system, brain or psychiatric disorders.
7. HIV infection with laboratory or clinical diagnosis.
8. Previous history of hepatitis C, chronic hepatitis B infection, or evidence of active hepatitis. Laboratory tests at the screening stage indicate seropositivity for hepatitis C or hepatitis B seropositivity (HBsAg positive). In addition, if HBsAg is negative but HBcAb is positive (regardless of HBsAb status), HBV DNA testing is required, and if positive, the subject should be excluded.
9. During the screening period, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase were more than 1.5 times of the upper limit of normal value, serum creatinine and bilirubin were more than 1.2 times of the upper limit of normal value, and serum albumin was less than 10% of the lower limit of normal value.
10. Bone marrow biopsy results within 6 months before enrollment showed that myelofibrosis score MF≥2.
11. There is a history of abnormal platelet aggregation that may affect the reliability of platelet count measurements.
12. Any medical history or condition that the investigator deems unsuitable for participation in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-05-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Treatment response | From the start of study treatment (Day 1) up to the end of week 4, week 8 and week 12.
  Number of participants achieving a platelet count >=30×10^9/L and at least doubling of the baseline count at Week 4, Week 8, and Week 12.

SECONDARY OUTCOMES:
Long-term treatment response | From the start of study treatment (Day 1) up to the end of week 24.
  The proportion of subjects who achieve efficacy (R) at 24weeks of treatment.
Withdrawal of eltrombopag | From the start of study treatment (Day 1) up to the end of week 24.
  The proportion of subjects who successfully stop TPO-RAs within 24 weeks.
Drug efficacy 1 | From the start of study treatment (Day 1) up to the end of week 4, week 8, week 12 and week 24.
  Number of participants achieving a platelet count >=30×10^9/L at week 4, week 8, week 12 and week 24 in ITP patients with or without positive autoantibody.
Time to Response | From the start of study treatment (Day 1) up to the end of week 24.
  The time required from the start of treatment to the first time a subject's platelet count was greater than or equal to 30×109/L and at least a two-fold increase from the baseline platelet count.
Duration of response | From the start of study treatment (Day 1) up to the end of week 24.
  Total duration of subject's platelet count ≥30×109/L
Drug efficacy 2 | From the start of study treatment (Day 1) up to the end of week 4, week 8, week 12 and week 24.
  Number of participants achieving a platelet count >=50×10^9/L at week 4, week 8, week 12 and week 24
emergency treatment | From the start of study treatment (Day 1) up to the end of week 24.
  The proportion of subjects receiving emergency treatment
Evaluation of effectiveness | From the start of study treatment (Day 1) up to the end of week 24.
  Number of participants that reduced or discontinued baseline concomitant ITP medications during the whole 24 weeks.
Number of participants with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale. | From the start of study treatment (Day 1) up to the end of week 24.
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Number of participants with clinically significant bleeding as assessed using the bleeding scale for pediatric patients with ITP. | From the start of study treatment (Day 1) up to the end of week 24.
  The bleeding scale for pediatric patients with ITP is a measure of bleeding severity with the following grades: Grade 1 (minor) Minor bleeding, few petechiae (≤100 total) and/or ≤5 small bruises (≤3 cm in diameter), no mucosal bleeding；Grade 2 (mild) Mild bleeding, many petechiae (>100 total) and/or >5 large bruises (>3 cm in diameter), no mucosal bleeding；Grade 3 (moderate) Moderate bleeding, overt mucosal bleeding, troublesome lifestyle；Grade 4 (severe) Severe bleeding, mucosal bleeding leading to decrease in Hb>2 g/dL or suspected internal hemorrhage；
Health-related quality of life survey of subjects(HRQoL)-1 | From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use ITP-PAQ (ITP Patient Assessment Questionnaire) to assess the HRQoL before and after treatment.
Health-related quality of life survey of subjects(HRQoL)-2 | From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use FACIT-F（functional assessment of chronic illness therapy- fatigue）to assess the HRQoL before and after treatment.
Health-related quality of life survey of subjects(HRQoL)-3 | From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use Kids' ITP tool KIT、to assess the HRQoL before and after treatment.
Health-related quality of life survey of subjects(HRQoL)-4 | From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use Pediatric Quality of Life Inventory PedsQL to assess the HRQoL before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D.,Ph.D, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neunert C, Terrell DR, Arnold DM, Buchanan G, Cines DB, Cooper N, Cuker A, Despotovic JM, George JN, Grace RF, Kuhne T, Kuter DJ, Lim W, McCrae KR, Pruitt B, Shimanek H, Vesely SK. American Society of Hematology 2019 guidelines for immune thrombocytopenia. Blood Adv. 2019 Dec 10;3(23):3829-3866. doi: 10.1182/bloodadvances.2019000966. PMID 31794604
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Result] Working Group of Chinese Guideline for the Diagnosis and Treatment of Childhood Primary Immune Thrombocytopenia; Subspecialty Group of Hematologic Diseases, the Society of Pediatrics, Chinese Medical Association; Editorial Board, Chinese Journal of Pediatrics. [Adapted guideline for the diagnosis and treatment of primary immune thrombocytopenia for Chinese children (2021)]. Zhonghua Er Ke Za Zhi. 2021 Oct 2;59(10):810-819. doi: 10.3760/cma.j.cn112140-20210509-00397. Chinese. PMID 34587675
- [Result] Cheng G, Saleh MN, Marcher C, Vasey S, Mayer B, Aivado M, Arning M, Stone NL, Bussel JB. Eltrombopag for management of chronic immune thrombocytopenia (RAISE): a 6-month, randomised, phase 3 study. Lancet. 2011 Jan 29;377(9763):393-402. doi: 10.1016/S0140-6736(10)60959-2. Epub 2010 Aug 23. PMID 20739054
- [Result] Wong RSM, Saleh MN, Khelif A, Salama A, Portella MSO, Burgess P, Bussel JB. Safety and efficacy of long-term treatment of chronic/persistent ITP with eltrombopag: final results of the EXTEND study. Blood. 2017 Dec 7;130(23):2527-2536. doi: 10.1182/blood-2017-04-748707. Epub 2017 Oct 17. PMID 29042367
- [Result] Yang R, Li J, Jin J, Huang M, Yu Z, Xu X, Zhang X, Hou M. Multicentre, randomised phase III study of the efficacy and safety of eltrombopag in Chinese patients with chronic immune thrombocytopenia. Br J Haematol. 2017 Jan;176(1):101-110. doi: 10.1111/bjh.14380. Epub 2016 Oct 13. PMID 27734464
- [Result] Cheng X, Fu L, Ma J, Gu H, Chen Z, Zhao L, Wang X, Wu R. Spotlight on eltrombopag in pediatric ITP in China: a long-term observational study in real-world practice. Blood Adv. 2021 Oct 12;5(19):3799-3806. doi: 10.1182/bloodadvances.2020004110. PMID 34605871
- [Result] Qu M, Zhou J, Yang SJ, Zhou ZP. Efficacy and safety of rituximab for minors with immune thrombocytopenia: a systematic review and meta-analysis. J Int Med Res. 2020 Oct;48(10):300060520962348. doi: 10.1177/0300060520962348. PMID 33115308
- [Result] Ayad N, Grace RF, Al-Samkari H. Thrombopoietin receptor agonists and rituximab for treatment of pediatric immune thrombocytopenia: A systematic review and meta-analysis of prospective clinical trials. Pediatr Blood Cancer. 2022 Mar;69(3):e29447. doi: 10.1002/pbc.29447. Epub 2021 Dec 28. PMID 34962697
- [Result] Sui T, Zhang L, Zhou ZP, Xue F, Ge J, Yang RC. [Efficacy and safety of two different low-dose rituximab regimens for Chinese adult patients with immune thrombocytopenia]. Zhonghua Xue Ye Xue Za Zhi. 2011 Sep;32(9):583-6. Chinese. PMID 22338149
- [Result] Liu X, Huang Y, Chen Y, Liu W, Xue F, Zhang L, Yang R. [Clinical analysis of lower doses rituximab for children primary immune thrombocytopenia]. Zhonghua Xue Ye Xue Za Zhi. 2014 Dec;35(12):1079-82. doi: 10.3760/cma.j.issn.0253-2727.2014.12.007. Chinese. PMID 25543701
- [Result] Provan D, Arnold DM, Bussel JB, Chong BH, Cooper N, Gernsheimer T, Ghanima W, Godeau B, Gonzalez-Lopez TJ, Grainger J, Hou M, Kruse C, McDonald V, Michel M, Newland AC, Pavord S, Rodeghiero F, Scully M, Tomiyama Y, Wong RS, Zaja F, Kuter DJ. Updated international consensus report on the investigation and management of primary immune thrombocytopenia. Blood Adv. 2019 Nov 26;3(22):3780-3817. doi: 10.1182/bloodadvances.2019000812. PMID 31770441
- [Result] Bussel JB, de Miguel PG, Despotovic JM, Grainger JD, Sevilla J, Blanchette VS, Krishnamurti L, Connor P, David M, Boayue KB, Matthews DC, Lambert MP, Marcello LM, Iyengar M, Chan GW, Chagin KD, Theodore D, Bailey CK, Bakshi KK. Eltrombopag for the treatment of children with persistent and chronic immune thrombocytopenia (PETIT): a randomised, multicentre, placebo-controlled study. Lancet Haematol. 2015 Aug;2(8):e315-25. doi: 10.1016/S2352-3026(15)00114-3. Epub 2015 Jul 28. PMID 26688484
- [Result] Grainger JD, Locatelli F, Chotsampancharoen T, Donyush E, Pongtanakul B, Komvilaisak P, Sosothikul D, Drelichman G, Sirachainan N, Holzhauer S, Lebedev V, Lemons R, Pospisilova D, Ramenghi U, Bussel JB, Bakshi KK, Iyengar M, Chan GW, Chagin KD, Theodore D, Marcello LM, Bailey CK. Eltrombopag for children with chronic immune thrombocytopenia (PETIT2): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Oct 24;386(10004):1649-58. doi: 10.1016/S0140-6736(15)61107-2. Epub 2015 Jul 28. PMID 26231455